CLINICAL TRIAL: NCT04917263
Title: IMMUNOlogical Microenvironment in REctal Adenocarcinoma Treatment. Predictors of Sustained Complete Response After Neoadjuvant Chemo/Radiotherapy for Locally Advanced Rectal Cancer
Brief Title: IMMUNOlogical Microenvironment in REctal Adenocarcinoma Treatment.
Acronym: IMMUNOREACT2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); Azienda Ospedaliera di Padova (Other); Istituto Oncologico Veneto IRCCS (Other); Azienda ULSS 3 Serenissima (Other); Azienda Ulss 2 Marca Trevigiana (Other)
Responsible Party: Sponsor
Other Study IDs: AIRC IG2019 23381 IMMUNOREACT2
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; complete response; neoadjuvant therapy; immune surveillance
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Mucosal samples from healthy tissue surrounding the cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective
  Interventions: Diagnostic Test: Immunohistochemistry, Flow citometry, Trascriptome analysis
- Prospective
  Interventions: Diagnostic Test: Immunohistochemistry, Flow citometry, Trascriptome analysis

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry, Flow citometry, Trascriptome analysis — we will perform immunohistochemistry, flow cytometry, transcriptomic analysis, mRNA microarray and mutational profiling

SUMMARY:
Background The current management on rectal cancer based on TNM staging has some limitations. In locally advanced rectal cancer after neoadjuvant therapy the persistence of a complete response to therapy cannot be accurately predicted by the simple tumor regression grade. The current guidelines recommend the complete rectal resection with a total mesorectal excision. The implications for patients' quality of life are evident even in case of sphincter sparing surgery. Moreover, in both cases the cancer sample available for the analysis can be small or inexistent. Hypothesis The main hypothesis underlying our research is that the aggressiveness of rectal cancer is determined by the complex interactions between the malignant cells and their immune microenvironment. The second hypothesis is that relevant trace of this cross talk between tumor cells and immune microenvironment can be detected in the normal mucosa surrounding the cancer according to the concept of field cancerization.

Aims The aim of this project is to analyze the healthy rectal mucosa surrounding the cancer to identify traces of immunosurveillance mechanisms and of field cancerization and to use them to obtain a composite prognostic test to predict recurrence after complete response at neoadjuvant therapy in case of locally advanced rectal cancer.

Experimental Design This prognostic test will be constructed on the combinatory analysis of the transcriptome, immune and epithelial cells cross-talk, immune checkpoints and miRNA expression in normal rectal mucosa surrounding cancer. The project aim is to identify, among locally advanced rectal cancer, those with sustained complete response to neoadjuvant chemo/radiotherapy. The study is articulated in two steps. In step A, we will retrospectively analyze archival tissue samples in order to identify the most performing biomarkers; in step B, we will validate the prognostic performance of the markers identified in phase I through a prospective analysis of rectal mucosa specimen.

DETAILED DESCRIPTION:
Locally advanced rectal cancer: which treatment after complete response after neoadjuvant therapy? Combined treatment for locally advanced rectal cancer achieves a 5-year overall survival close to90% [15]. This multimodal approach can be also applied to elderly patients with stage III rectal cancer obtaining improved oncological outcomes [16]. Some patients with rectal cancer who receive neoadjuvant chemoradiotherapy (nCRT) achieve a pathologic complete response (pCR) and may be eligible for less radical surgery or non-operative management [17]. Moreover, complete regression of the rectal cancer after neoadjuvant chemoradiation therapy have been confirmed by clinical and radiographic evaluation-this is known as complete clinical response (cCR). The "watch and wait" approach was first proposed by Dr. Angelita Habr-Gama in Brazil in 2009. Those patients with cCR are followed with rigorousphysical, endoscopical, and imaging surveillance [18]. Several studies aimed to identify variables that predict pCR after nCRT for rectal cancer. A large retrospective review of the NCDB performed from 2006 to 2011, including a total of 23,747 patients identified the clinical factors associated with pCR. They were lower tumor grade, lower clinical T and N stage, higher radiation dose, and delaying surgery by more than 6-8weeks after the end of radiation, while lack of health insurance was linked with a lower likelihood of pCR [17]. Another study identified predictive factors in the models included tumor length, tumor circumferential extent, age, and ApoA1 [19]. A different study showed that responders after neoadjuvant chemoradiation had a lower incidence of cytokeratin 20 positive circulating tumor cells compared to non-responders, which might be a result of effective systemic and local treatment prior to surgery [20]. Finally, the role of immune microenvironment was investigated analyzing Foxp3(+), CD3(+), CD4(+), CD8(+) and IL-17(+) cell density in post-CRT surgical samples from 128 patients with rectal cancer. Stromal Foxp3(+) cell density was strongly associated with tumor regression grade. A low stromal Foxp3(+) cell density was observed in 84% of patients who had a pathologic complete response (pCR) compared to41% of patients who did not. Low stromal Foxp3(+) cell density was also associated with improved recurrence-free survival. Regulatory T cells in the tumor microenvironment may inhibit response to neoadjuvant CRT and may represent a therapeutic target in rectal cancer [21].

Hypotheses and Specific aims The main hypothesis underlying our research is that aggressiveness of rectal cancer is determined by the complex interactions between the malignant cells and the local immune microenvironment. Our hypothesis is that the local immune activation may involve the "healthy" rectal mucosa surrounding the cancer and the sampling of this mucosa may provide useful information about rectal cancer behavior. In fact, a combination of different factors, including molecular signaling networks (i.e. checkpoint genes) within different cell population, presence of soluble chemical factors and quantity/quality of immune cells infiltrate will decide rectal cancer behavior and its response to neoadjuvant chemoradiation. Moreover, tumor cells actively interact with the microenvironment secreting and degrading extracellular matrix components, and the release of soluble molecules (e.g. miRNA) can significantly influence the inflammatory and immune responses of the "healthy" rectal mucosa surrounding the cancer. By using state of the art histological/molecular/immunological markers and bio-statistical analysis tools we aim to identify clinically relevant molecular targets to design effective therapeutic strategies for rectal cancer patients.

Therefore, the aim of the study is to identify a prognostic test that accurately predicts rectal cancer behavior even in case when the tumor samples are scarce (due to small size of early rectal cancer) or absent (in case of complete response to therapy). This prognostic test will be constructed on the combinatory analysis of the transcriptome, immune cells activation and checkpoints, epithelial cells activity as antigen presenting cells and miRNA expression in normal tissue specimens of prospectively collected rectal cancers. The question is how to identify, among locally advanced rectal cancer, those with immediate and sustained complete response to neoadjuvant chemo/radiotherapy. These patients might safely avoid a low rectal resection with all the consequences for their quality of life. In patients with locally advanced rectal cancer (N+) an ideal biomarker should be able to identify the cohort of patients that will have a complete response to neoadjuvant therapy and will not require further treatments.

Study design Tissue samples will be obtained from cancer tissue (if possible) and from normal rectal mucosa adjacent to the cancer at surgery. The very large number of patients need to answer the two questions imply a multicentric design. Complete medical record and follow-up will be collected from each center. The analysis will be centralized mostly in Azienda Ospedaliera di Padova. The study will be articulated in two parts each of them aiming to answer to one of the above described questions. Each part of the study will be articulated in a retrospective and exploratory step (A) and in a prospective validation step (B).

ELIGIBILITY:
Inclusion Criteria:

1. locally advanced (cT3-4 and/or N+, TNM stage II-III) low and medium rectal cancer (<11 cm) or low rectum adenocarcinoma cT≤2, at risk for abdominoperineal amputation, undergoing neoadjuvant therapy will be included in the study group.
2. Only neoadjuvant therapy protocols including long course radiotherapy (45 Gy) and fluoropyrimidine-based regimens will be included while short radiation therapy of radiation therapy or chemotherapy alone will be excluded
3. at least 6 weeks after the end of the neoadjuvant therapy will be included
4. Full availability of clinical records at least 1 year of follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to analyze 66 patients with pathological complete response and 66 patients without complete response after neoadjuvant therapy for locally advanced rectal cancer. Given an expected proportion of 20% of patients with complete response, we estimate to enroll a total number of 66/0.20=330 patients with early rectal cancer. However, we will performed flow cytometry, transcriptomic analysis, mRNA microarray and mutational profiling only in 132 patients (66 patients with complete response and 66 patients without complete response) in order to test the non-inferiority of AUC.
  Taking into account a 15-20% of locally advanced rectal cancer patients with pathological complete response to neoadjuvant therapy and a maximum of 7 prognostic factors (including markers and clinical factors) in the model, we aim to enroll 412 patients in this part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response on the operative specimen | first post operative month
  pathological complete response to neoadjuvant chemo/radiotherapy in locally advanced rectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Marco Scarpa, MD, PhD, Principal Investigator — Clinica Chirurgica I, Azienda Ospedale Università di Padova
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Italy

REFERENCES:
- [Derived] Becherucci G, Ruffolo C, Scarpa M, Scognamiglio F, Stepanyan A, Maretto I, Kotsafti A, De Simoni O, Pilati P, Franzato B, Scapinello A, Bergamo F, Massani M, Stecca T, Pozza A, Cataldo I, Brignola S, Pellegrini V, Fassan M, Guzzardo V, Dal Santo L, Salmaso R, Carlotta C, Dei Tos AP, Angriman I, Spolverato G, Chiminazzo V, Negro S, Vignotto C, Marchegiani F, Facci L, Rivella G, Bao QR, Baldo A, Pucciarelli S, Zizzo M, Businello G, Salmaso B, Parini D, Pirozzolo G, Recordare A, Tagliente G, Bordignon G, Merenda R, Licia L, Pozza G, Godina M, Mondi I, Verdi D, Da Lio C, Guerriero S, Piccioli A, Portale G, Zuin M, Cipollari C, Noaro G, Cola R, Candioli S, Gavagna L, Ricagna F, Ortenzi M, Guerrieri M, Tomassi M, Tedeschi U, Marinelli L, Barbareschi M, Bertalot G, Brolese A, Ceccarini L, Antoniutti M, Porzionato A, Agostini M, Cavallin F, Tussardi G, Di Camillo B, Bardini R, Castagliuolo I, Scarpa M. IMMUNOREACT 8: Immune markers of local tumor spread in patients undergoing transanal excision for clinically N0 rectal cancer. Surgery. 2025 Feb;178:108902. doi: 10.1016/j.surg.2024.09.043. Epub 2024 Nov 20. PMID 39572264